CLINICAL TRIAL: NCT04564742
Title: A Registry-based, Randomised, Double-blind, Placebo-Controlled Cardiovascular Outcomes Trial to Evaluate the Effect of Dapagliflozin on Cardiometabolic Outcomes in Patients Without Diabetes With Acute Myocardial Infarction at Increased Risk for Subsequent Development of Heart Failure
Brief Title: Dapagliflozin Effects on Cardiometabolic Outcomes in Patients With an Acute Heart Attack.
Acronym: DAPA-MI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D169DC00001; 2020-000664-31 (EudraCT Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-25 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Myocardial Infarction; Cardiovascular Outcome Trial
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental): Patients will be randomized 1:1 to either dapagliflozin or placebo
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo matching dapagliflozin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg tablets given once daily, per oral use
  Other Names: Forxiga TM; Farxiga TM
  Arms: Dapagliflozin
Drug: Placebo — Placebo matching dapagliflozin 10 mg tablets given once daily, per oral use
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of dapagliflozin versus placebo, given once daily in addition to Standard of Care (SoC) therapies for patients with myocardial infarction (MI), for hospitalisation for heart failure (HHF), cardiovascular (CV) death, and other cardiometabolic outcomes.

DETAILED DESCRIPTION:
This is a multicentre, parallel group double-blind, placebo-controlled phase 3 registry-based randomised controlled trial (R-RCT) in patients without diabetes presenting with myocardial infarction (MI) (ST segment elevation myocardial infarction (STEMI) or non-ST segment elevation myocardial infarction (NSTEMI)) and evidence of impaired regional or global LV systolic function or definite evidence of Q wave MI on ECG. In the study the effect of dapagliflozin versus placebo, given once daily in addition to SoC therapy will be evaluated for the hospitalisation for HF, CV death, and other cardiometabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 at the time of signing the informed consent
* Confirmed MI, either STEMI or NSTEMI, according to the fourth universal definition of MI (Thygesen et al 2019), within the preceding 7 days, or 10 days if earlier randomisation is not feasible
* Evidence of impaired regional or global LV systolic function at any timepoint during current MI-related hospitalisation (established with echocardiogram, radionuclide ventriculogram, contrast angiography or cardiac MRI) or definitive evidence on ECG of Q wave MI (defined as presence of Q waves in two or more contiguous leads, excluding leads III and aVR, and meeting all the following criteria: at least 1.5 mm in depth; at least 30 ms in duration; and, if R wave present, more than 25% of the size of the subsequent R wave)
* Hemodynamically stable at randomization (no episodes of symptomatic hypotension, or arrhythmia with haemodynamic compromise in the last 24 hours).
* Male or female
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
* Provision of signed and dated, written informed consent prior to any mandatory study specific procedures, sampling, and analyses

Exclusion Criteria:

* Known type 1 diabetes mellitus (T1DM) or T2DM at the time for admission. Patients with hyperglycaemia, but without a diagnosis of diabetes mellitus prior to the index event, are eligible at the discretion of the Investigator. Patients who present with signs and symptoms consistent with ketoacidosis, including nausea, vomiting, abdominal pain, malaise and shortness of breath should be assessed for ketoacidosis, and if ketoacidosis is confirmed the patient should not be randomized.
* Chronic symptomatic HF with a prior HHF within the last year and known reduced ejection fraction (LVEF≤40 %), documented before the current MI hospitalization
* Severe (eGFR <20 mL/min/1.73 m2 by local laboratory), unstable or rapidly progressing renal disease at the time of randomization
* Severe hepatic impairment (Child-Pugh class C) at the time of inclusion into the trial
* Active malignancy requiring treatment at the time of screening, except for basal cell- or squamous cell carcinoma of the skin, presumed possible to treat successfully
* Any non-CV condition, eg malignancy, with a life expectancy of less than two years based on the investigator´s clinical judgement
* Currently on treatment, or with an indication for treatment, with a sodium glucose co-transporter 2 inhibitor (SGLT2-inhibitor)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4017 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan James, Principal Investigator — Uppsala University; Jonas Oldgren, Study Chair — Uppsala University
Locations (93):
- Sweden (34):
  - Research Site, Alingsås
  - Research Site, Borås
  - Research Site, Eskilstuna
  - Research Site, Falun
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Halmstad
  - Research Site, Hässleholm
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Kalix
  - Research Site, Karlshamn
  - Research Site, Karlskoga
  - Research Site, Karlskrona
  - Research Site, Karlstad
  - Research Site, Kiruna
  - Research Site, Köping
  - Research Site, Lidköping
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Mölndal
  - Research Site, Norrköping
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Skellefteå
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Varberg
  - Research Site, Värnamo
  - Research Site, Västerås
  - Research Site, Ystad
- United Kingdom (59):
  - Research Site, Aberdeen
  - Research Site, Ashford
  - Research Site, Basingstoke
  - Research Site, Bath
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Bridgend
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Buckhurst Hill
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Clydebank
  - Research Site, Coventry
  - Research Site, Derby
  - Research Site, Dundee
  - Research Site, East Kilbride
  - Research Site, Edgbaston
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Gillingham
  - Research Site, Glasgow
  - Research Site, Harefield
  - Research Site, Harrow
  - Research Site, Headington
  - Research Site, Hull
  - Research Site, Kettering
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Lincoln
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Merthyr Tydfil
  - Research Site, Middlesbrough
  - Research Site, Newcastle upon Tyne
  - Research Site, Newport
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Pont-y-clun
  - Research Site, Portsmouth
  - Research Site, Rhyl
  - Research Site, Scarborough
  - Research Site, Sheffield
  - Research Site, Southampton
  - Research Site, Stevenage
  - Research Site, Stoke-on-Trent
  - Research Site, Sunderland
  - Research Site, Swansea
  - Research Site, Taunton
  - Research Site, Torquay
  - Research Site, Truro
  - Research Site, Wakefield
  - Research Site, Wigan
  - Research Site, Wolverhampton
  - Research Site, Worcester
  - Research Site, Worthing

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] James S, Erlinge D, Storey RF, McGuire DK, de Belder M, Eriksson N, Andersen K, Austin D, Arefalk G, Carrick D, Hofmann R, Hoole SP, Jones DA, Lee K, Tygesen H, Johansson PA, Langkilde AM, Ridderstrale W, Parvaresh Rizi E, Deanfield J, Oldgren J. Dapagliflozin in Myocardial Infarction without Diabetes or Heart Failure. NEJM Evid. 2024 Feb;3(2):EVIDoa2300286. doi: 10.1056/EVIDoa2300286. Epub 2023 Nov 11. PMID 38320489
- [Derived] James S, Erlinge D, Storey RF, McGuire DK, de Belder M, Bjorkgren I, Johansson PA, Langkilde AM, Ridderstrale W, Parvaresh Rizi E, Deanfield J, Oldgren J. Rationale and design of the DAPA-MI trial: Dapagliflozin in patients without diabetes mellitus with acute myocardial infarction. Am Heart J. 2023 Dec;266:188-197. doi: 10.1016/j.ahj.2023.08.008. Epub 2023 Aug 28. PMID 37648579
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169DC00001&attachmentIdentifier=6a26fd8c-8a16-4e88-be06-fe8f77ed02d1&fileName=D169DC00001_Final_Protocol_Redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169DC00001&attachmentIdentifier=e44ba4b4-00be-45a8-b7a0-d42b1e24a19d&fileName=D169DC00001_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169DC00001&attachmentIdentifier=b1e72f98-98f3-46d8-9ff9-cb04417bbf85&fileName=D169DC00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapa 10 mg: Active, Green, plain, diamond shaped, film coated tablet, 10 mg once daily
- Placebo: Control, Green, plain, diamond shaped, film coated tablets, once daily
Period: Overall Study
Arm/Group | Dapa 10 mg | Placebo
Started | 2019 | 1998
Completed | 2014 | 1994
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Consent Withdrawal | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa 10 mg | Placebo | Total
Number analyzed (Participants) | 2019 | 1998 | 4017
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (Years) | 63.0 (11.06) | 62.8 (10.64) | 62.9 (10.85)
Age, Customized [Number; unit: Participants]
  >65 years | 831 | 799 | 1630
  <=65 years | 1188 | 1199 | 2387
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The full analysis set population
  Participants
    Female | 388 | 419 | 807
    Male | 1631 | 1579 | 3210
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The full analysis set population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 64 | 52 | 116
    Black or African American | 8 | 15 | 23
    Native Hawaiian or other Pacific Islander | 0 | 0 | 0
    Other | 40 | 37 | 77
    White | 1905 | 1893 | 3798
    MISSING | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Analysis of the Hierarchical Primary Composite Endpoint (Full Analysis Set)
Description: Study participants received dapagliflozin 10 mg or matching placebo, given once daily in addition to SoC. Overall, the mean study duration was 12.0 months (time in study until last visit) with an accumulated 4023.9 participant-years. The maximum study duration for any participant was 29 months.
  "Number of Events" for NYHA corresponds to the number of participants with a non-missing value for NYHA functional class at the last visit, and that all participants with a non-missing value take part in the analysis comparing their NYHA class value with all other participants with a NYHA value, according to the win-ratio method.
Time Frame: 29 months
Population: All participants are included in the analysis; Each row item displays the number of participants for the given event, and without preceding events defined in the hierarchical order.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2019 | 1998
Participants
  The hierachical composite endpoint of all components | 1990 | 1970
  Death, adjudicated | 41 | 33
  Hospitalisation due to HF | 32 | 41
  Non-fatal MI | 29 | 32
  AF/Flutter event | 8 | 15
  New onset of T2DM | 40 | 74
  NYHA Classification at last visit, measuring limitations of physical activity | 1839 | 1773
  Body Weight decrease of at least 5% at last visit | 684 | 468
Statistical Analysis 1: Comparison: Dapa 10 mg vs Placebo; The primary objective of the study was to determine if the clinical benefit of dapagliflozin was superior as compared with placebo, utilizing a hierarchical composite endpoint and win-ratio (WR) method. With a presumed WR of 1.20, 4000 patients were provide an 80% statistical power for the primary endpoint, maintaining a 1:1 allocation between treatments. The primary analysis was based on the intention-to-treat principle using the Full Analysis Set; Test type: Superiority; p < 0.001, Win Ratio Analysis — A closed testing procedure including a pre-specified hierarchical ordering of the primary and secondary endpoints was utilised. No multiplicity control was placed on the exploratory endpoints; Win Ratio (WR) = 1.34, 95% CI 2-sided [1.20 to 1.50]

ADVERSE EVENTS:
Time Frame: Time frame was from date of randomization and up to and including last day in study, up to 29 months.
Groups:
- Dapa 10 mg; Placebo: Description (Arm-group)
Arm/Group | Dapa 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 41/2019 | 33/1998
Serious Adverse Events (participants affected / at risk) | 449/2019 | 404/1998
Other Adverse Events (participants affected / at risk) | 0/2019 | 0/1998
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=2019) | Placebo (N=1998)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 16 (16) | 24 (24)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 39 (43) | 30 (34)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 2 (2)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 8 (8)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Primary biliary cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 36 (39) | 36 (40)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 3 (3)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 33 (35) | 32 (34)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fascial infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 20 (21) | 17 (21)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 10 (11) | 5 (5)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Parapharyngeal space infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 22 (24) | 15 (16)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 3 (4)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9) | 7 (7)
Urosepsis (Infections and infestations) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 2 (2) | 1 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery dissection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 18 (21)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (5)
Atrial flutter (Cardiac disorders) | 5 (5) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 7 (7) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5) | 8 (8)
Large intestine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm papilla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 40 (55) | 39 (43)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 4 (4)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 9 (9)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 3 (3) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 14 (14) | 10 (10)
Transient ischaemic attack (Nervous system disorders) | 4 (5) | 4 (4)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 14 (15) | 16 (16)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (8) | 2 (2)
Cardiac pseudoaneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 2 (2)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cardiac sarcoidosis (Cardiac disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (9)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 7 (7) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Elective procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 3 (3)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 9 (10) | 8 (8)
Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhage coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 4 (4)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 11 (11) | 5 (5)
Postinfarction angina (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (5) | 4 (5)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 5 (5)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 5 (5)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 5 (5)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT04564742/Prot_004.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT04564742/SAP_005.pdf